CLINICAL TRIAL: NCT07080073
Title: Comparative Effects of Maitland and Mulligan Spinal Mobilizations Along With Canal Enlargement Exercises in Patients of Lumbar Spinal Stenosis
Brief Title: Effects of Maitland and Mulligan Spinal Mobilizations Along With Canal Enlargement Exercises in Lumbar Spinal Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0166 Areej
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Spinal Stenosis; Low Back Pain
Keywords: Manual Therapy; Canal Enlargement Exercises; Pain; Disability
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland Mobilization Group (Experimental): Participants in this group will receive Maitland Grade III central posterior-anterior spinal mobilizations targeting the lumbar spine. The intervention will be administered by a licensed physiotherapist with the patient in a prone position, applying oscillatory mobilization for 3 sets of 40 seconds with 1-minute rest intervals. This will be combined with:
  Interventions: Other: Maitland Mobilization Group
- Mulligan Mobilization Group (Experimental): Participants in this group will receive Mulligan spinal mobilizations with lower limb movement (SNAGs). The therapist will apply sustained passive glides to the lumbar spinous process while the patient actively elevates the leg in a pain-free range. Mobilizations will be performed in 3 sets of 7-10 repetitions. This will be combined with:
  Interventions: Other: Mulligan Mobilization Group

INTERVENTIONS:
Other: Maitland Mobilization Group — Participants in this group will receive Maitland Grade III central posterior-anterior spinal mobilizations targeting the lumbar spine. The intervention will be administered by a licensed physiotherapist with the patient in a prone position, applying oscillatory mobilization for 3 sets of 40 seconds with 1-minute rest intervals.
  Canal enlargement exercises (bilateral knee-to-chest, LION stretch, cat-camel exercise) The total treatment will be administered four sessions per week for three weeks (12 sessions total).
  Arms: Maitland Mobilization Group
Other: Mulligan Mobilization Group — Participants in this group will receive Mulligan spinal mobilizations with lower limb movement (SNAGs). The therapist will apply sustained passive glides to the lumbar spinous process while the patient actively elevates the leg in a pain-free range. Mobilizations will be performed in 3 sets of 7-10 repetitions.
  Canal enlargement exercises (bilateral knee-to-chest, LION stretch, cat-camel exercise) The total treatment will be administered four sessions per week for three weeks (12 sessions total).
  Arms: Mulligan Mobilization Group

SUMMARY:
This randomised controlled trial will evaluate the comparative effects of Maitland versus Mulligan spinal mobilization techniques, when combined with canal enlargement exercises, in patients with lumbar spinal stenosis (LSS). A total of 38 participants aged 25-40 years with confirmed unilateral LSS will be randomly assigned to receive either Maitland mobilizations or Mulligan mobilizations, along with standard physiotherapy and canal enlargement exercises. The intervention will be administered over three weeks, with four sessions per week. Primary outcomes will include pain intensity (measured by Numeric Pain Rating Scale), disability (Modified Oswestry Disability Index), and symptom severity (Swiss Spinal Stenosis Score), assessed at baseline and post-treatment. This study aims to inform physiotherapy practice by identifying the more effective manual therapy technique for improving functional outcomes in LSS.

DETAILED DESCRIPTION:
This single-blinded, randomised controlled trial is designed to compare the effects of two manual therapy techniques, Maitland central posterior-anterior Grade III mobilizations and Mulligan spinal mobilizations (SNAGs), when combined with canal enlargement exercises and conventional physiotherapy. Thirty-eight participants with confirmed unilateral lumbar spinal stenosis will be recruited from the outpatient physiotherapy department at Allama Iqbal Memorial Teaching Hospital, Sialkot.

Participants will be randomly assigned to one of two intervention groups using sealed opaque envelopes. Group A will receive Maitland mobilizations in addition to canal enlargement exercises and conventional physiotherapy, while Group B will receive Mulligan mobilizations along with the same exercise and conventional therapy protocol. The intervention will be administered four times per week over a period of three weeks (total of 12 sessions).

The canal enlargement protocol includes bilateral knee-to-chest exercises, LION stretches, and cat-camel movements, all of which aim to increase lumbar flexion and spinal canal space. Conventional physiotherapy treatment will include the application of hot packs, transcutaneous electrical nerve stimulation (TENS), and stretching of the hamstrings and piriformis muscles.

Primary outcomes will be assessed at baseline and after the 3-week intervention. These include:

Pain intensity (Numeric Pain Rating Scale, NPRS)

Functional disability (Modified Oswestry Disability Index, MODI)

Symptom severity (Swiss Spinal Stenosis Score, SSSS)

Data will be analysed using appropriate parametric and non-parametric statistical tests, based on data distribution. The findings of this study will provide insight into which mobilization technique is more effective in reducing pain and disability and improving function in patients with lumbar spinal stenosis. This may contribute to the development of more evidence-based physiotherapy protocols for LSS management.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 25-40 years

  * Both males and females will be included
  * Patient with low back pain along with unilateral radiating symptoms
  * Having symptoms from at least 3 months with pain severity not more than 7 on NPRS
  * Diagnosed case of slipped disc or herniation causing spinal stenosis, confirmed by physical examination and/or MRI.

Exclusion Criteria:

* Chronic inflammatory or infectious disease, neoplasm, hematological disorders, traumatic vertebral injuries, Spondylitis

  * Any concurrent major disease like renal failure, diabetes, cancer, tumor.
  * Low back pain with bilateral radiating symptoms.
  * Pregnancy
  * Cognitive alteration and non-co-operative patient
  * Spinal surgery

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline and at the end of 3 weeks (post-intervention)
  Pain will be assessed using the 11-point Numeric Pain Rating Scale (NPRS), where 0 represents "no pain" and 10 represents "worst possible pain." The scale is a reliable self-reported tool for evaluating pain intensity in musculoskeletal conditions.
Modified Oswestry Disability Index (MODI) | Baseline and at 3 weeks post-intervention
  Functional disability will be assessed using the Modified Oswestry Disability Index (MODI), a validated questionnaire that measures the degree of disability related to low back pain. Scores range from 0% (no disability) to 100% (maximum disability).
Swiss Spinal Stenosis Score (SSSS) | Baseline and at 3 weeks post-intervention
  The Swiss Spinal Stenosis Score (SSSS) will be used to assess symptom severity and physical function specific to lumbar spinal stenosis. The tool includes subscales for symptom intensity and function, with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Zia, Phd Scholar, Principal Investigator — Riphah International University; Areej Ijaz, MSc Student, Principal Investigator — Riphah International University
Locations (1):
- Allama Iqbal memorial teaching hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munakomi S, Foris LA, Varacallo MA. Spinal Stenosis and Neurogenic Claudication. 2023 Aug 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK430872/ PMID 28613622
- [Background] Homayouni K, Naseri M, Zaravar F, Zaravar L, Karimian H. Comparison of the Effect of Aquatic Physical Therapy and Conventional Physical Therapy in Patients with Lumbar Spinal Stenosis (a Randomized Controlled Trial). Journal of Musculoskeletal Research. 2015;18(01)
- [Background] Gaur P, Goyal M, Singh G. Manual therapy and canal enlargement exercises versus conventional physiotherapy in lumbar stenosis - a study protocol. Revista Pesquisa em Fisioterapia. 2021;11
- [Background] Kumar S, A N. Effect of Integrated Exercise Protocol in Lumbar Spinal Stenosis as Compare with Conventional Physiotherapy- A Randomized Control Trial. International Journal of Neurorehabilitation. 2017;04(06).
- [Background] Maitland G. Management of lumbar spine disorder. Maitland's vertebral manipulation 8th ed United Kingdom: Churchill Livingstone. 2013:230-6.